CLINICAL TRIAL: NCT00002845
Title: TREATMENT OF METASTATIC MELANOMA WITH RECOMBINANT INTERLEUKIN-2
Brief Title: Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Blumenthal Cancer Center at Carolinas Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065084; CMC-09-95-16B; NCI-V96-1037
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells.

PURPOSE: Phase II trial to study the effectiveness of interleukin-2 in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response and survival rates of patients with metastatic melanoma following induction with high-dose and maintenance with low-dose interleukin-2. II. Assess the toxicity of this regimen.

OUTLINE: All patients receive high-dose interleukin-2 over 24 hours, followed by low-dose interleukin-2 for 4 days in the absence of toxicity. Patients receive a second cycle beginning 9-13 days after completion of the first cycle, with response assessed approximately 2 months after initiating therapy. Patients with stable or responding disease receive a second course as above; those with a continued response may receive additional courses provided toxicity is limited. Patients are followed for survival.

PROJECTED ACCRUAL: 20 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven melanoma that is metastatic No tumor replacement of 25% or more of liver on CT or MRI No involvement of the CNS or a major nerve Measurable disease required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80%-100% Life expectancy: More than 3 months Hematopoietic: No coagulopathy (i.e., platelets less than 80,000) Hepatic: Bilirubin normal Renal: Creatinine normal Cardiovascular: No abnormal cardiac stress test in patients over 50 years of age or with possible cardiac disease suggested by history, physical exam, or EKG Pulmonary: FEV1 or VC greater than 65% of predicted in patients with significant smoking history or with suspected pulmonary disease by history, physical exam, or x-ray Other: No site of ongoing bleeding No systemic infection No HIV antibody No HBsAg No requirement for steroids No psychiatric disease that precludes informed consent or protocol treatment No second malignancy except: Basal cell skin carcinoma Carcinoma in situ of the cervix No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: No prior interleukin-2 At least 28 days since treatment for melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1995-09

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. White, MD, Study Chair — Blumenthal Cancer Center at Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States